CLINICAL TRIAL: NCT01140490
Title: Sub-total Parathyroidectomy Reduces Vascular Calcification in Haemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Guangdong General Hospital, Department of nephrology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8020
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2009-01

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Sub-total Parathyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sub-total Parathyroidectomy (No Intervention)
  Interventions: Procedure: Sub-total Parathyroidectomy

INTERVENTIONS:
Procedure: Sub-total Parathyroidectomy — Sub-total Parathyroidectomy

SUMMARY:
The aim of this study was to evaluate whether successful sub-total parathyroidectomy retards cardiovascular calcification in patients with hemodialysis and to investigate the mechanism .

DETAILED DESCRIPTION:
Hyperparathyroidism (PHPT) in patients with end-stage renal disease have been shown to have an increased morbidity and mortality mainly due to cardiovascular disease. The precise mechanism of cardiovascular disease in PHPT is not well understood . The excess in cardiovascular mortality is significantly and independently related to serum calcium, the connection between the biochemical disturbances and the cardiovascular disorders in PHPT patients is not necessarily a cause-and-effect relationship. Indeed, the impact of surgical cure of hyperparathyroidism on cardiovascular risk factors and mortality is controversial. Some studies suggest that cardiovascular risk markers remained unaltered after Sub-total Parathyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* The patients receiving hemodialysis treatment, with elevated intact parathyroid hormone (iPTH) levels > 800pg/ml on two or more occasions.
* Patients with parathyroid nodular or diffuse hyperplasia identified by ultrasound imaging or radioisotope scan.

Exclusion Criteria:

* Patients with significant background valvular heart disease
* Patients who are unfit for general anaesthesia
* Patients with acute myocardial infarction within recent two months
* Patients with poor general condition
* Patients with plans for living related kidney transplant within 1 year
* Patients with previous history of parathyroidectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in vascular calcium scores | 12 months

SECONDARY OUTCOMES:
Change in left ventricular systolic and diastolic function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shi wei, MD PHD, Principal Investigator — Chinese Nephrology Committee
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China